CLINICAL TRIAL: NCT03007472
Title: Clinical Evaluation of the Cochlear Nucleus(R) CI532 Cochlear Implant in Adults
Brief Title: Clinical Evaluation of the Cochlear Nucleus CI532 Cochlear Implant in Adults
Acronym: SME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cochlear (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLTD5685
Record Dates: First submitted 2016-12-27; First posted 2017-01-02 (Estimated); Results first posted 2020-12-03 (Actual); Last update posted 2020-12-30 (Actual); Status verified 2020-12

CONDITIONS: Hearing Loss, Sensorineural
Keywords: cochlear implant, sound processor
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- CI532/N7 study group (Experimental): All subjects will receive a CI532 cochlear implant (intervention) and be fit with the CP1000 sound processor
  Interventions: Device: CI532; Device: Nucleus 7

INTERVENTIONS:
Device: CI532 — Cochlear implant
  Other Names: Slim Modiolar Electrode; 532
Device: Nucleus 7 — Sound processor
  Other Names: N7; CP1000

SUMMARY:
The purpose of this study is to gather long-term data on the FDA approved CI532 cochlear implant, and CP1000 (Nucleus 7) sound processor

DETAILED DESCRIPTION:
Appropriate candidates will receive a CI532 cochlear implant and be fit with the CP1000 sound processor. Imaging will be completed pre-op, intra-op, and post-op to assess implant location. Speech perception testing as well as subjective questionnaires will be administered over 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Adults 18 years or older who have a bilateral postlinguistic sensorineural hearing loss.
2. Limited benefit from amplification as defined by test scores of 40% correct or less in the ear to be implanted and 50% or less in the contralateral ear on a recorded monosyllabic word test I. Consistent with the Minimum Speech Test Battery (2011), it is required that all subjects be evaluated at 60 dBA presentation level.
3. Bilateral moderate sloping to profound hearing loss
4. Minimum of 30 days experience with appropriately fit bilateral amplification, fit using the standardized National Acoustics Laboratory (NAL) fitting method
5. Proficient in English
6. Ability to complete testing -

Exclusion Criteria:

1. Previous cochlear implantation
2. Pre-linguistically deafened (onset of hearing loss at less than two years of age)
3. Ossification or any other cochlear anomaly that might prevent complete insertion of the electrode array
4. Duration of severe to profound hearing loss greater than 20 years
5. Diagnosis of retro-cochlear pathology
6. Diagnosis of auditory neuropathy
7. Unrealistic expectations on the part of the subject regarding the possible benefits, risks, and limitations that are inherent to the surgical procedure and use of the prosthetic device
8. Unwillingness or inability to comply with all investigational requirements
9. Additional cognitive, medical or social handicaps that would prevent completion of all study requirements-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2017-02-15 (Actual); Primary Completion 2018-12-03 (Actual); Study Completion 2020-03-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jillian Crosson, PhD, Study Director — Senior Manager of Clinical Services; Megan Mears, AuD, Study Director — Clinical Project Manager
Locations (10):
- United States (10):
  - Rocky Mountain Ear Center, Englewood, Colorado
  - University of Iowa, Iowa City, Iowa
  - University of Michigan, Ann Arbor, Michigan
  - The Center for Hearing and Balance Disorders, Chesterfield, Missouri
  - Midwest Ear Institute, Kansas City, Missouri
  - Washington University, St Louis, Missouri
  - New York University, New York, New York
  - The Ohio State University, Columbus, Ohio
  - Hearts for Hearing, Oklahoma City, Oklahoma
  - Dallas Ear Institute, Dallas, Texas

REFERENCES:
- [Background] Grutters JP, Joore MA, van der Horst F, Verschuure H, Dreschler WA, Anteunis LJ. Choosing between measures: comparison of EQ-5D, HUI2 and HUI3 in persons with hearing complaints. Qual Life Res. 2007 Oct;16(8):1439-49. doi: 10.1007/s11136-007-9237-x. Epub 2007 Jul 24. PMID 17647093
- [Background] Hiller W, Goebel G. Factors influencing tinnitus loudness and annoyance. Arch Otolaryngol Head Neck Surg. 2006 Dec;132(12):1323-30. doi: 10.1001/archotol.132.12.1323. PMID 17178943
- [Background] Meinert,C(1986).ClinicalTrials:Design,Conduct,andAnalysis.OxfordUniversityPress,NewYork.
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Background] PETERSON GE, LEHISTE I. Revised CNC lists for auditory tests. J Speech Hear Disord. 1962 Feb;27:62-70. doi: 10.1044/jshd.2701.62. No abstract available. PMID 14485785
- [Background] Spahr AJ, Dorman MF, Litvak LM, Van Wie S, Gifford RH, Loizou PC, Loiselle LM, Oakes T, Cook S. Development and validation of the AzBio sentence lists. Ear Hear. 2012 Jan-Feb;33(1):112-7. doi: 10.1097/AUD.0b013e31822c2549. PMID 21829134
- [Derived] Kelsall D, Lupo J, Biever A. Longitudinal outcomes of cochlear implantation and bimodal hearing in a large group of adults: A multicenter clinical study. Am J Otolaryngol. 2021 Jan-Feb;42(1):102773. doi: 10.1016/j.amjoto.2020.102773. Epub 2020 Oct 22. PMID 33161258
- [Derived] Wick CC, Kallogjeri D, McJunkin JL, Durakovic N, Holden LK, Herzog JA, Firszt JB, Buchman CA; CI532 Study Group. Hearing and Quality-of-Life Outcomes After Cochlear Implantation in Adult Hearing Aid Users 65 Years or Older: A Secondary Analysis of a Nonrandomized Clinical Trial. JAMA Otolaryngol Head Neck Surg. 2020 Oct 1;146(10):925-932. doi: 10.1001/jamaoto.2020.1585. PMID 32857114
- [Derived] Buchman CA, Herzog JA, McJunkin JL, Wick CC, Durakovic N, Firszt JB, Kallogjeri D; CI532 Study Group. Assessment of Speech Understanding After Cochlear Implantation in Adult Hearing Aid Users: A Nonrandomized Controlled Trial. JAMA Otolaryngol Head Neck Surg. 2020 Oct 1;146(10):916-924. doi: 10.1001/jamaoto.2020.1584. PMID 32857113

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CI532/N7 Study Group
Started | 96
Completed | 91
Not Completed | 5
Not completed — Did not have aidable contralateral thresholds at the time | 2
Not completed — Death | 2
Not completed — Loss to Follow Up | 1

BASELINE CHARACTERISTICS:
Arm/Group | CI532/N7 Study Group
Number analyzed (Participants) | 96
Age, Continuous [Mean (Full Range); unit: years] | 67.39 [23 to 91]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 62
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 96
Ipsilateral Ear Mean - Duration of Hearing Loss [Mean (Standard Deviation); unit: years] | 21.7 (14)
Contralateral Ear Mean - Duration of Hearing Loss [Mean (Standard Deviation); unit: years] | 26.7 (14)

OUTCOME MEASURES:

1. Primary Outcome: Change From Pre- to 6 Months Post-implantation Speech Recognition in Quiet in the Implanted Ear Alone
Description: Group mean Consonant Nucleus Consonant (CNC) word recognition in quiet measured pre-operatively and again at 6 month post sound processor activation compared to the group mean score in the preoperative, best unilateral condition. The CNC word test has a score range of 0-100% with higher values indicating better scores.
Time Frame: Preoperatively and 6 months post sound processor activation
Measure: Mean (Standard Deviation); unit: percentage of correct words
Arm/Group | CI532/N7 Study Group
Number analyzed (Participants) | 96
percentage of correct words
  Baseline Ipsilateral Aided | 14.6 (11.6)
  6 Month CI/Best Unilateral | 60.9 (21.09)

2. Secondary Outcome: Evaluation of Change in Pre and Post Implantation Speech Recognition in Noise Scores in the Implanted Ear Alone
Description: Group mean AzBio sentence in noise score in the best unilateral condition compared to the group mean score in the preoperative, unilateral aided condition. The AzBio sentence test has a score range of 0-100% with higher values indicating better scores.
Time Frame: Preoperatively and 6 months post sound processor activation
Measure: Mean (Standard Deviation); unit: percentage of correct AzBio sentences
Arm/Group | CI532/N7 Study Group
Number analyzed (Participants) | 96
percentage of correct AzBio sentences
  Baseline Ipsilateral Aided +10 SNR | 14.8 (17.24)
  6 Month CI/Best Unilateral +10 SNR | 42.7 (26.21)

3. Secondary Outcome: Change in Pre and Post Implantation Score on the Health Utility Index-3 (HUI3)
Description: Group mean HUI3 score post sound processor activation compared to the scores measured preoperatively. The HUI3 consists of eight attributes of general health (vision, hearing, speech, mobility, dexterity, emotion, cognition, and pain) with five or six levels per attribute. For each respondent, health status is described as a vector that combines the levels of each attribute. This information is then converted into a utility score of HRQL on a scale from perfect health (1.0) to death (0).
Time Frame: Preoperatively and 6 months post sound processor activaton
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CI532/N7 Study Group
Number analyzed (Participants) | 94
score on a scale
  Baseline | 0.46 (0.2)
  6 Month | 0.64 (0.197)

4. Other Pre Specified Outcome: Frequency Specific Thresholds and Speech Recognition in Noise or Quiet
Description: Frequency-specific thresholds at standard audiometric frequencies for each ear, and speech recognition in quiet (CNC words) or noise (AzBio sentences) in best unilateral and/or electric alone.
Time Frame: 12 months post-activation
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Speech Perception in Quiet and Noise With Change in Cochlear Implant Programming
Description: Two optional study visits to evaluate whether a change in cochlear implant programming, specifically an increase in the number of channels will improve subject speech perception in quiet and noise.
Time Frame: Following 12-month study visit but prior to 36-month interval.
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | CI532/N7 Study Group
All-Cause Mortality (participants affected / at risk) | 2/96
Serious Adverse Events (participants affected / at risk) | 16/96
Other Adverse Events (participants affected / at risk) | 26/96
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CI532/N7 Study Group (N=96)
Acid Reflux (Gastrointestinal disorders) | 1 (1)
Active Meniere's Disease/Vertigo (Ear and labyrinth disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Atrial Fibrillation requiring Ablation Procedure (Cardiac disorders) | 1 (1)
CI Explanted Due to Non-Auditory Stimulation (Product Issues) | 1 (1)
Coxsackievirus, subsequent labyrinthitis/vestibular neuritis (Ear and labyrinth disorders) | 1 (1)
CVA (cerebrovascular accident) (Vascular disorders) | 1 (1)
Cardio-respiratory failure (Cardiac disorders) | 1 (1) — Death secondary to cardio-respiratory failure, presistent tachycardia secondary to myotonic distrophy, stage Y3 N0 colon carcinoma, sepsis, VRE, acidosis
Alcoholic cirrhosis of the liver (Hepatobiliary disorders) | 1 (1) — Death-complications
Decreased Hearing in Non-Implanted Ear (Ear and labyrinth disorders) | 1 (1)
Dehydration (General disorders) | 1 (1)
Diagnosed with prostate cancer (Reproductive system and breast disorders) | 1 (1)
Electrode Tip Foldover (Injury, poisoning and procedural complications) | 1 (1)
Heart Attack (Cardiac disorders) | 1 (2)
Seizure (Nervous system disorders) | 1 (1)
TIA/Stroke (Vascular disorders) | 1 (1)
Tip Rollover (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CI532/N7 Study Group (N=96)
Dizziness (General disorders) | 14 (14)
Vertigo (Ear and labyrinth disorders) | 13 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-06-28): https://cdn.clinicaltrials.gov/large-docs/72/NCT03007472/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-04): https://cdn.clinicaltrials.gov/large-docs/72/NCT03007472/SAP_001.pdf